CLINICAL TRIAL: NCT01207375
Title: Improving New Learning in Traumatic Brain Injury: A Randomized Clinical Trial
Brief Title: Improving New Learning and Memory in Traumatic Brain Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kessler Foundation (Other)
Collaborators: U.S. Department of Education (U.S. Federal Agency)
Responsible Party: Principal Investigator, Nancy Chiaravalloti, Director, Neuropsychology & Neuroscience Lab, Kessler Foundation
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ndcnidrr2007
Record Dates: First submitted 2010-09-21; First posted 2010-09-22 (Estimated); Last update posted 2015-04-03 (Estimated); Status verified 2015-04

CONDITIONS: Traumatic Brain Injury
Keywords: memory; learning; Traumatic Brain Injury; cognition; treatment; therapy
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- experimental group (Experimental): The experimental group will receive memory retraining exercises administered on a laptop computer twice a week for 5 weeks (10 training sessions).
  Interventions: Behavioral: memory retraining exercises
- Placebo control group (Placebo Comparator): The placebo control group will receive placebo memory exercises administered on a laptop computer twice a week for five weeks (10 placebo control sessions).
  Interventions: Behavioral: placebo control memory exercises

INTERVENTIONS:
Behavioral: memory retraining exercises — Memory retraining exercises will be administered on a laptop computer twice a week for 5 weeks (10 training sessions).
  Arms: experimental group
Behavioral: placebo control memory exercises — Placebo control memory exercises will be administered on a laptop computer twice a week for five weeks (10 placebo control sessions.
  Arms: Placebo control group

SUMMARY:
The current study is a double-blind, placebo-control randomized clinical trial examining the efficacy of memory retraining in Traumatic Brain Injury (TBI). Impairment in higher level cognitive processing, such as new learning and memory, is one of the most common deficits in individuals with TBI and such deficits have been shown to exert significant negative impact on multiple aspects of everyday life, including occupational and social functioning. Despite these findings, few studies have attempted to treat these cognitive deficits in order to improve the everyday functioning of individuals with TBI. The current proposal will evaluate (a)the efficacy of this treatment protocol within a TBI population,(b) the impact of the treatment on everyday functioning, (c) the long term efficacy of the treatment and (c) the utility of booster sessions in facilitating long-term treatment effects. The investigators will randomly assign individuals with TBI, with documented impairment in new learning abilities, to a memory retraining group or a placebo control group. Both groups will undergo baseline, immediate and long-term follow-up assessment consisting of: (1) a traditional neuropsychological battery and (2) an assessment of global functioning examining the impact of the treatment on daily activities. This design will allow us to evaluate the efficacy of this particular memory retraining technique in a TBI population through the assessment of cognitive function via a standard evaluation. In addition, the investigators will be able to draw conclusions regarding the impact of this particular memory remediation program on everyday life from questionnaires completed by the participant and a significant other. Optional enrollment in pre/post neuroimaging will also allow us to look at changes in the brain.

DETAILED DESCRIPTION:
Impairments in higher level cognitive processing, such as new learning and memory, are among the most common deficits in individuals with Traumatic Brain Injury (TBI) and such deficits have been shown to exert significant negative impact on multiple aspects of everyday life, including occupational and social functioning. Despite these findings, few studies have attempted to remediate these cognitive deficits in order to improve the everyday functioning of individuals with TBI

Therefore, we will conduct a double-blind, placebo-controlled, randomized clinical trial, applying a memory rehabilitation technique to a large sample of TBI participants. This protocol has been well-validated with other neurological populations and preliminary evidence in support of its use in MS now exists. Individuals with TBI, with documented impairment in memory and new learning, will be randomly assigned to either a memory retraining group or a placebo control group. Outcome will be measured through two mechanisms: (1) a traditional neuropsychological (NP) battery and (2) an assessment of global functioning (AGF) examining the impact of the treatment on daily activities. Both groups will undergo baseline, immediate follow-up, and long-term follow-up assessments consisting of a traditional NP evaluation, which examines objective performance on well-validated measures of cognitive function, and an AGF, which includes self-report measures of memory abilities, self-efficacy, quality of life, and occupational functioning. In this way, we will be able to objectively evaluate the presence or absence of changes in memory performance through a NP assessment, while also evaluating the impact of this treatment protocol on an individual's everyday life through the AGF. While most studies evaluating the efficacy of cognitive retraining usually employ a pre-training and post-training evaluation, such evaluations have been criticized for their lack of ecological validity. The present design allows the assessment of the efficacy of this particular memory retraining technique within an TBI population using traditional measures, as well as the assessment of the impact that such a rehabilitation technique has on everyday life. In addition, we will include a 6-month follow-up assessment to measure the long-term impact of this treatment on objective cognitive functioning, through a NP assessment, and everyday life, through an AGF. Finally, half of the participants in the experimental group will participate in monthly "booster sessions" following the completion of treatment and we will evaluate the impact of these sessions on the maintenance of treatment effects over time. A subset of the sample will also complete pre and post neuroimaging to evaluate changes in cerebral activation.

The documentation of the efficacy of memory retraining in TBI, particularly on everyday functioning, could have a significant impact on symptom management and quality of life in the lives of persons. As such, specific aims of the current research protocol are as follows.

Aim 1. This study will objectively evaluate the clinical utility of a memory retraining protocol to improve performance on objective tests of new learning and memory in a large sample of individuals with TBI with documented deficits in this area.

Aim 2. We will increase the generalizability and real life application of assessment techniques by assessing outcome following cognitive retraining with more global measures of everyday life. An objective measure of everyday functioning will be included, as well as numerous subjective measures of everyday functioning, which will be gathered via established self-report instruments, as well as ratings by a significant other.

Aim 3: This study will evaluate the long-term efficacy of this memory retraining protocol through the inclusion of a 6-month follow-up assessment. Many cognitive remediation studies in the literature examine the efficacy of the treatment immediately following program completion. However, given the time, expense, and labor involved in such intensive treatment, it is important to demonstrate the long-term efficacy of such a program. The current study therefore goes beyond the typical protocol length to evaluate the long-term impact such treatment will have on objective testing and on an individual's daily life.

Aim 4: We will examine the need for and impact of "booster sessions" following the completion of treatment. "Booster sessions" have been shown to be efficacious in maximizing the long term benefit of cognitive retraining in research with other populations. However, the utility of booster sessions in a TBI population has never been investigated.

ELIGIBILITY:
Inclusion Criteria:

* English as primary language
* Diagnosis of TBI, at least one year post-injury

Exclusion Criteria:

* ages less than 18 or greater than 59
* previous head injury, stroke, seizures, or any other significant neurological history
* Medications: persons on steroids, benzodiazepines, and/or neuroleptics will not be included
* Individuals with an active diagnosis of Major Depressive Disorder, Schizophrenia, Bipolar Disorder I or II will be excluded from the study
* Significant history of drug or alcohol abuse
* Poor Visual Acuity (corrected vision in worse eye < 20/60), diplopia, or nystagmus
* Inability to understand directions and following one, two, and three step commands
* Intact New Learning and Memory: Only individuals that show impaired performance on a memory test will be included in the study

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2008-01; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Scores on memory tests | Three points in time: pre-treatment, immediately following treatment and 6 months after treatment is completed

SECONDARY OUTCOMES:
Reports of emotional functioning, memory functioning and quality of life | Three points in time: pre-treatment, immediately following treatment and 6 months after treatment is completed

CONTACTS AND LOCATIONS:
Overall Officials: Nancy D Chiaravalloti, Ph.D., Principal Investigator — Kessler Foundation
Locations (1):
- Kessler Foundation Research Center, West Orange, New Jersey, United States